CLINICAL TRIAL: NCT00902746
Title: Phase3, Open-Label, Long-Term, NSAID-Add-on, Clinical Trial of NPC-01 for Treatment of Dysmenorrhea Associated With Endometriosis.
Brief Title: Efficacy and Safety, Long-Term Study of NPC-01 to Treat Dysmenorrhea Associated With Endometriosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nobelpharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC-01-1
Record Dates: First submitted 2009-05-07; First posted 2009-05-15 (Estimated); Results first posted 2014-06-13 (Estimated); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NPC-01 (Experimental): Norethisterone, Ethinyl Estradiol
  Interventions: Drug: NPC-01

INTERVENTIONS:
Drug: NPC-01 — This study consist of the following steps.
  Step 1(Norethisterone 0.6mg, Ethinyl Estradiol 0.035mg):From first study medication to 3th menstrual cycles.
  Step 2(Norethisterone 1mg, Ethinyl Estradiol 0.035mg):
  After interim analysis of the results of step 1, in the case of the efficacy results meet prespecified criterion, same dose level will be continued to 13th menstrual cycles including step 1. If the results do not meet prespecified criterion, the dose will be increased to Norethisterone 1mg, Ethinyl Estradiol 0.035mg and be continued newly until 13th menstrual cycle from this point.

SUMMARY:
The purpose of this long-term study is to determine whether NPC-01 is effective in the treatment of dysmenorrhea associated with endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Dysmenorrhea associated with endometriosis

Exclusion Criteria:

* Severe hepatopathy
* Pregnant woman

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2009-05; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naoki Terakawa, M.D.,Ph.D., Study Director — Nissay Hospital,Osaka,Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total 168 patients were consented and registered at minus 2 cycles of study drug administration as provisional registration.
  After provisional registration, investigators confirmed their eligibility of patients by test gynecological examination, transvaginal ultrasound etc.) and 149 patients were formally registered for this study.
Groups:
- NPC-01: Norethisterone, Ethinyl Estradiol
  NPC-01: This study consist of the following steps.
  Step 1(Norethisterone 0.6mg, Ethinyl Estradiol 0.035mg):From first study medication to 3th menstrual cycles.
  Step 2(Norethisterone 1mg, Ethinyl Estradiol 0.035mg):
  After interim analysis of the results of step 1, in the case of the efficacy results meet prespecified criterion, same dose level will be continued to 13th menstrual cycles including step 1. If the results do not meet prespecified criterion, the dose will be increased to Norethisterone 1mg, Ethinyl Estradiol 0.035mg and be continued newly until 13th menstrual cycle from this point.
Period: Overall Study
Arm/Group | NPC-01
Started | 149
Initiation of Study Drug Administration | 148
Transfer to Step 2 | 133
Completed | 113
Not Completed | 36
Not completed — Protocol Violation | 7
Not completed — Withdrawal by Subject | 16
Not completed — Adverse Event | 8
Not completed — Lost to Follow-up | 3
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Population: Baseline analysis were carried out on 147 patients except 1 patients who has no available data of efficacy and safety in 148 cases that study drug administration was started.
Groups:
- NPC-01: Norethisterone, Ethinyl Estradiol
  NPC-01: This study consist of the following steps.
  Step 1(Norethisterone 0.6mg, Ethinyl Estradiol 0.035mg):From first study medication to 3th menstrual cycles.
  Step 2(Norethisterone 0.6mg, Ethinyl Estradiol 0.035mg, or Norethisterone 1mg, Ethinyl Estradiol 0.035mg):
  After interim analysis of the results of step 1, in the case of the efficacy results meet prespecified criterion, same dose level will be continued to 13th menstrual cycles including step 1. If the results do not meet prespecified criterion, the dose will be increased to Norethisterone 1mg, Ethinyl Estradiol 0.035mg and be continued newly until 13th menstrual cycle from this point.
Arm/Group | NPC-01
Number analyzed (Participants) | 147
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (7.12)
Age, Customized [Number; unit: participants]
  Under 30 years of age | 51
  30 year of age and older | 96
Sex/Gender, Customized [Number; unit: participants]
  Female | 147
Total Dysmenorrhea Score (VRS; Verbal Rating Scale) [Mean (Standard Deviation); unit: units on a scale] | 4.1 (0.99)
Visual Analogue Scale [Mean (Standard Deviation); unit: units on a scale] | 53.1 (21.49)

OUTCOME MEASURES:

1. Primary Outcome: Patient Response to Treatment for Dysmenorrhea, as Evaluated by Difference of Total Dysmenorrhea Score (Baseline/Pretreatment-End of Treatment)
Description: The detail of dysmenorrhea score that was used in this study is the following. These subscales summed for a total dysmenorrhea score (minimum 0 to maximum 6). Pain score None 0 : None Mild 1 : There are some troubles for work Moderate 2 : Needing to rest in bed and/or affecting work Severe 3 : Morre than 1 day in bed and not possible to work
  Drug score (during a menstrual period) None 0 : None Mild 1 : taking analgesics for 1 days Moderate 2 : taking analgesics for 2 days Severe 3 : taking analgesics more than 3 days
Time Frame: 52 weeks
Population: This analysis was carried out for 112 patients whom end of study data was available on FAS.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NPC-01
Number analyzed (Participants) | 112
units on a scale | 2.4 (1.80)

2. Secondary Outcome: Difference in the Visual Analog Scale (VAS) of Dysmenorrhea (Baseline/Pretreatment-dnd of Treatment)
Description: VAS stands for Visual Analogue Scale of pain. The scale was rated as a graphic rating scale. as a 100mm baseline from 0:No pain to 100:Worst possible pain.
Time Frame: 52 weeks
Population: This analysis was carried out for 112 patients whom end of study data was available on FAS.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NPC-01
Number analyzed (Participants) | 112
units on a scale | 28.4 (25.13)

ADVERSE EVENTS:
Time Frame: From study administration to 15 cycles of menstruation, an average of 14 months
Arm/Group | NPC-01
Serious Adverse Events (participants affected / at risk) | 5/147
Other Adverse Events (participants affected / at risk) | 147/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NPC-01 (N=147)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 1 (1)
Cellulitis orbital (Infections and infestations) | 1 (1)
Haemorrhagic ovrian cyst (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NPC-01 (N=147)
Abdominal discomfort (Gastrointestinal disorders) | 11 (20)
Abdominal pain upper (Gastrointestinal disorders) | 17 (29)
Constipation (Gastrointestinal disorders) | 10 (10)
Dental caries (Gastrointestinal disorders) | 12 (13)
Diarrhoea (Gastrointestinal disorders) | 14 (34)
Gastritis (Gastrointestinal disorders) | 9 (9)
Nausea (Gastrointestinal disorders) | 25 (42)
Malaise (General disorders) | 13 (17)
Cystitis (Infections and infestations) | 9 (9)
Gastroenteritis (Infections and infestations) | 13 (14)
Influenza (Infections and infestations) | 12 (12)
Nasopharyngitis (Infections and infestations) | 95 (242)
Blood triglycerides increased (Investigations) | 9 (11)
Weight increased (Investigations) | 10 (10)
Protein urine present (Investigations) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (13)
Headache (Nervous system disorders) | 53 (220)
Amenorrhoea (Reproductive system and breast disorders) | 10 (11)
Hypomenorrhoea (Reproductive system and breast disorders) | 22 (27)
Menorrhagia (Reproductive system and breast disorders) | 24 (42)
Metrorrhagia (Reproductive system and breast disorders) | 132 (916)
Oligomenorrhoea (Reproductive system and breast disorders) | 67 (135)
Polymenorrhoea (Reproductive system and breast disorders) | 19 (29)
Breast discomfort (Reproductive system and breast disorders) | 8 (11)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 14 (14)
Acnes (Skin and subcutaneous tissue disorders) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between the sponsor and PI that no restricts the PI's right but need to discuss the timing of publish date of trial results after the trial is completed.